CLINICAL TRIAL: NCT03462797
Title: Opioid Physiology Project
Acronym: OPP
Status: Completed | Type: Observational
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: 17-05380-XP
Record Dates: First submitted 2017-10-24; First posted 2018-03-13 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Tolerance; Withdrawal; Addiction; Epigenetic Changes
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The coordinator will collect saliva samples (ORG-500) from study subjects at the start of study and at follow up visits. Saliva samples will be collected non-invasively using the DNA Oragene sample collection kits (http://www.dnagenotek.com). The investigator will then perform genome-wide DNA methylation assay using the Illumina Infinium MethylationEPIC array (https://www.illumina.com). The investigator will monitor the longitudinal change in the methylome that may be induced by short-term opioid use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current project seeks to explore the use of emergent biosensor technology to detect opioid use. The investigators goal is to recruit 60 opioid naïve patients presenting at the College of Dentistry at UTHSC. Candidate participants must be scheduled for an upcoming dental procedure that will involve subsequent pain management using oral opioid medication. Participants will be consented prior to any study procedures. All participant information from this study will be kept strictly confidential (e.g., no individual data will be shared with the College of Dentistry).

DETAILED DESCRIPTION:
Opioid overdose is a leading cause of accidental death in the USA, with death rates rising steadily over the last 20 years (CDC, 2015). Of the over 22,000 deaths relating to pharmaceutical overdose in 2011, three quarters involved opioid analgesics (Fletcher et al., 2011). Increases in problematic opioid use have paralleled a corresponding increase in drug treatment admissions (DOHH, 2014). Drug treatment programs currently focus on behavioral and pharmacologic interventions to sustain abstinence, and success is typically measured by self-reports or urine drug screening (NIDA, 2016). Both measurement methods are limited by such factors as recall bias, distortion, and lack of precision (Fishman et al., 2000). A detection method that accurately detects opioid use as it occurs in real time would provide several distinct advantages, including the ability to obtain environmental and behavioral contexts surrounding relapse as well as an opportunity for targeted interventions.

The current project seeks to explore the use of emergent biosensor technology to detect opioid use. The investigators goal is to recruit 60 opioid naïve patients presenting at the College of Dentistry at UTHSC. Candidate participants must be scheduled for an upcoming dental procedure that will involve subsequent pain management using oral opioid medication. Participants will be consented prior to any study procedures. All participant information from this study will be kept strictly confidential (e.g., no individual data will be shared with the College of Dentistry).

Participants who are enrolled will complete baseline questionnaires regarding psychological and behavioral risks of substance use. Next, participants will be asked to wear the wristband sensor for 1 day prior to surgery, and up to 30 days post-surgery, or as long as opioid medication is prescribed. Physiological measurement will be conducted via the Empatica E4 wristband biosensor, which measures electrodermal activity, skin temperature, and locomotion data. Opioid use will detected through biosensor activity. Participants will be recruited over a 6 month period, in cohorts of 10. All study procedures will be approved by the UTHSC IRB.

Hilbert transform analyses combined with paired t-tests will be used to compare the biosensor data: (A) within subjects, before and after administration of opioids; and (B) between subjects, controlling for hand dominance, gender, and length of prescription.

Results of analyses will be shared with the College of Dentistry, and will subsequently be disseminated through a peer-reviewed publication.

Role of the College of Dentistry:

* To refer patients to Karen Derefinko's study team for possible recruitment into the study prior to the scheduled surgery.
* If possible, to allow a research coordinator to consent and interview participants on site in an available private room.
* To provide prescription data (type, dose, and duration) to study team, with signed participant consent.

Epigenetics:

Environmental exposures including prescription drugs and drugs of abuse can have a pronounce effect on the epigenome (Nestler, 2014; Nielsen et al., 2012). There is growing evidence that use of opioids results in changes in DNA methylation, an important epigenetic modification that can alter gene expression. Such changes may play a mechanistic role in forming an "epigenetic memory" of drug exposure and development of dependence (Doehring et al., 2013; Tuesta & Zhang, 2014). For this study, the coordinator will collect buccal swabs (cheek epithelial cells) from study subjects at the start of study and at follow up visits. Buccal cells will be collected non-invasively using the DNA Genotek sample collection kits (http://www.dnagenotek.com). The investigator will then perform genome-wide DNA methylation assay using the Illumina Infinium MethylationEPIC array (https://www.illumina.com). The investigator will evaluate the longitudinal change in the methylome that may be induced by short-term opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 or over)
* Opioid naive
* Getting a dental surgery where clinicians will prescribe opioid medication
* Ability to consent
* English as primary language
* Willingness to wear biosensor
* Willingness to complete daily log
* Willingness to provide saliva samples (epigenetics)

Exclusion Criteria:

* Inability to wear biosensor
* Other cause of pain (that may lead to other opioid use)
* Current drug or alcohol depend
* Inability to Consent
* Pregnancy
* Incarceration
* Musculoskeletal causes of pain limiting motion
* Upper Extremity Amputation
* Individuals with Developmental Disabilities

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Our study population will be recruited for the University of Tennessee College of Dentistry. Recruited populations will be opioid naive individuals that are scheduled for an upcoming dental surgery that will result in an opioid medication be prescribed for pain management.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Physiological changes | Physiological activity recording will start 24 to 48 hours before dental surgery date. Physiological activity will be stopped 2 days after discontinuation of opioid self-administration and will not exceed 30 days from surgery date.
  We will be measuring physiological changes from pre- to post-opioid administration through the Empatica E4 electronic wristband. This device measures 5 physiological parameters:
  1. Physical activity through an accelerometer measuring movement on x,y, and z axes.
  2. Heart rate measured in beats per minute (BMP)
  3. Skin conductance measured in µs (microseconds)
  4. Temperature measured in Celsius (°C)
  5. Blood volume pulse measured in nm (nanometers)
  and DNA methylation after self administration of opioid medication.

SECONDARY OUTCOMES:
DNA Methlyation changes | Initial saliva sample will be collected before surgery date. Second sample will be collected 2 days after discontinuation of opioid self-administration. Last sample will be collected at the 30 days from surgery date.
  We will be measuring DNA methylation markers and their changes from pre- to post-opioid administration through Ilumina Infinium methylation EPIC. More specifically, we will be looking at changes in β-values, which are the ratio of (DNA methylation)/(DNA methylation + DNA unmethylation). We will use DNA Genotek's Oragene Discover for saliva collection.

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Derefinko, PhD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee College of Dentistry, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salgado Garcia FI, Indic P, Stapp J, Chintha KK, He Z, Brooks JH, Carreiro S, Derefinko KJ. Using wearable technology to detect prescription opioid self-administration. Pain. 2022 Feb 1;163(2):e357-e367. doi: 10.1097/j.pain.0000000000002375. PMID 34270522